CLINICAL TRIAL: NCT05735236
Title: Comparison of Methods in Post Operative Knee Arthroscopy Rehabilitation
Acronym: ACL BFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1052
Record Dates: First submitted 2023-01-18; First posted 2023-02-21 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): Participants undergo standard post-operative physical therapy as prescribed by their surgeon.
- BFR Cuff (Active Comparator): Patients undergo standard post-operative physical therapy as prescribed by their surgeon with the addition of a Blood Flow Restriction (BFR) cuff that is used during their exercises.
  Interventions: Device: BFR Cuff

INTERVENTIONS:
Device: BFR Cuff — The BFR cuff will be applied to the proximal thigh of the surgical leg while the patient completes specified physical therapy exercises.80% occlusion pressure will be determined by PT's in clinic through the use of a Delphi unit. Subjects will then be able to use the Saga Fitness app to adjust this pressure if it differs from the automatic calibrated pressure.
  Other Names: Blood Flow Restriction Device; Blood Flow Restriction Cuff
  Arms: BFR Cuff

SUMMARY:
The aim of this study is to investigate the efficacy of blood flow restriction (BFR) therapy in post-operative rehabilitation following knee arthroscopy for primary ACL reconstruction. BFR has been shown to effect time to return to activity and strength postoperatively. This study aims to analyze the effects of BFR therapy in patients who underwent primary ACL reconstruction surgery compared to controls. Participants will be randomized into either a treatment (BFR Cuff) or control (no BFR cuff) group. All participants will follow standard of care (SOC) physical therapy protocol for 12 weeks after surgery according to their treatment group. Strength and patient outcome measures will be recorded throughout the 2 year study period.

DETAILED DESCRIPTION:
The aim of this study is to investigate the efficacy of blood flow restriction (BFR) therapy in post operative rehabilitation following knee arthroscopy. The current standard of care and post-operative pain levels can limit patients from applying load necessary to increase muscle size and strength development due to partial weight baring after surgery. We hypothesize that immediate and consistent use of BFR augmenting our current standard post operative knee arthroscopy rehabilitation protocol will result in greater improvement in strength and quicker achievement of phase-based rehabilitation goals. We hypothesize that these objective improvements in strength will correlate with clinically meaningful improvement in Tegner activity scale, International Knee Documentation Committee (IKDC), return to sport, Lower Extremity Functional Scale (LEFS), pain and resiliency (patient reported outcome, PRO) scores indicative of greater functional recovery compared to our standard rehabilitation protocol alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary knee arthroscopy for ACL reconstruction without meniscus repair
* Completing initial 12 weeks of physical therapy at the Steadman Hawkins Clinic in Denver
* Patients with access to smartphone device

Exclusion Criteria:

* Bilateral knee surgeries to be performed within 12 weeks of each other
* Patients received meniscus repairs, chondral lesion repair/transplants,
* Prior surgery on the same knee
* Anyone who meets the following contraindications for BFR therapy:

  * Deep Vein Thrombosis (DVT)

    * Pulmonary Embolism
    * Hemorrhagic/Thrombolytic Stroke
    * Clotting Disorders
    * Hemophilia or taking blood thinners
    * Pregnant or up to 6 months post-partum
    * Untreated Hypertension
    * Untreated Hypotension
    * Rhabdomyolysis or recent traumatic injury

      2. Exclusion criteria will be evaluated via the medical record as well as by the expert opinion of the physician.

      3. If at any point in the study a subject develops one of the above contraindications, they will be removed from the study.

      4. If a subject becomes pregnant while participating in the intervention portion of the study, they will be removed.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Knee extensor strength | 6 months
  Strength of knee extensors via handheld dynamometry (HHD) and reported as a measure of limb symmetry index (LSI) comparing operative limb to non-operative lim

SECONDARY OUTCOMES:
hamstrings musculature strength | 6 months
  Strength of knee flexors via handheld dynamometry (HHD) and reported as a measure of limb symmetry index (LSI) comparing operative limb to non-operative limb.
single leg squat test | 6 months
  Performance on a Repeated Single Leg Squat test to 45 deg knee flexion over the course of 90 seconds reported as a measure of LSI
Tegner Activity Scale | 6 months
  Tegner Activity Scale: Range 0 (disability because of knee problems) - 10 (national or international level soccer)
LEFS | 2 years
  Range 0 (extreme difficulty) -100 (nodifficulty);MDIC = Δ 123
Pain NPRS | 2 Years
  Range 1 (low pain) -10 (high pain); MDC = Δ 34
PROMIS Pain | 2 Years
  Range 0 (low pain) -100 (highpain); MDC = Δ 85
PROMIS Physical Function | 2 Years
  Range 0 (low function) -100 (high function); MDC = Δ 85
Brief Resiliency Score (BRS) | 2 Years
  Range 1(low resilience) -5 (high resilience); MDC = Δ low (1-2.99) to normal (3-4.3) to high (4.31-5)
ACL-RSI | 2 Years
  Range 1 (low function) -100 (high function); MDC = ∆15.1 for short form version
IKDC | 2 Years
  Range 1 (low function) -100 (high function); MDC = ∆8.8 low to ∆15.6 high

CONTACTS AND LOCATIONS:
Overall Officials: James Genuario, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UCHealth Steadman Hawkins Clinic, Centennial, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Proximal, Distal, and Contralateral Effects of Blood Flow Restriction Training on the Lower Extremities: A Randomized Controlled Trial. Sports Health. 2019 Mar/Apr;11(2):149-156. doi: 10.1177/1941738118821929. Epub 2019 Jan 14. PMID 30638439
- [Result] Tabata S, Suzuki Y, Azuma K, Matsumoto H. Rhabdomyolysis After Performing Blood Flow Restriction Training: A Case Report. J Strength Cond Res. 2016 Jul;30(7):2064-8. doi: 10.1519/JSC.0000000000001295. PMID 26677831
- [Result] Slysz J, Stultz J, Burr JF. The efficacy of blood flow restricted exercise: A systematic review & meta-analysis. J Sci Med Sport. 2016 Aug;19(8):669-75. doi: 10.1016/j.jsams.2015.09.005. Epub 2015 Sep 28. PMID 26463594
- [Result] Yasuda T, Fukumura K, Fukuda T, Uchida Y, Iida H, Meguro M, Sato Y, Yamasoba T, Nakajima T. Muscle size and arterial stiffness after blood flow-restricted low-intensity resistance training in older adults. Scand J Med Sci Sports. 2014 Oct;24(5):799-806. doi: 10.1111/sms.12087. Epub 2013 Jun 3. PMID 23730848
- [Result] Charles D, White R, Reyes C, Palmer D. A SYSTEMATIC REVIEW OF THE EFFECTS OF BLOOD FLOW RESTRICTION TRAINING ON QUADRICEPS MUSCLE ATROPHY AND CIRCUMFERENCE POST ACL RECONSTRUCTION. Int J Sports Phys Ther. 2020 Dec;15(6):882-891. doi: 10.26603/ijspt20200882. PMID 33344004
- [Result] Hung M, Saltzman CL, Kendall R, Bounsanga J, Voss MW, Lawrence B, Spiker R, Brodke D. What Are the MCIDs for PROMIS, NDI, and ODI Instruments Among Patients With Spinal Conditions? Clin Orthop Relat Res. 2018 Oct;476(10):2027-2036. doi: 10.1097/CORR.0000000000000419. PMID 30179950
- [Result] Grzybowski JS, Malloy P, Stegemann C, Bush-Joseph C, Harris JD, Nho SJ. Rehabilitation Following Hip Arthroscopy - A Systematic Review. Front Surg. 2015 May 26;2:21. doi: 10.3389/fsurg.2015.00021. eCollection 2015. PMID 26075208
- [Result] Chahal J, Van Thiel GS, Mather RC 3rd, Lee S, Song SH, Davis AM, Salata M, Nho SJ. The Patient Acceptable Symptomatic State for the Modified Harris Hip Score and Hip Outcome Score Among Patients Undergoing Surgical Treatment for Femoroacetabular Impingement. Am J Sports Med. 2015 Aug;43(8):1844-9. doi: 10.1177/0363546515587739. Epub 2015 Jun 15. PMID 26078452
- [Result] Bronner S, Chodock E, Urbano IER, Smith T. Psychometric Properties of the Dance Functional Outcome Survey (DFOS): Reliability, Validity, and Responsiveness. J Orthop Sports Phys Ther. 2019 Feb;49(2):64-79. doi: 10.2519/jospt.2019.8247. Epub 2018 Jul 27. PMID 30053790
- [Result] Enseki K, Harris-Hayes M, White DM, Cibulka MT, Woehrle J, Fagerson TL, Clohisy JC; Orthopaedic Section of the American Physical Therapy Association. Nonarthritic hip joint pain. J Orthop Sports Phys Ther. 2014 Jun;44(6):A1-32. doi: 10.2519/jospt.2014.0302. PMID 24881906
- [Result] Luebbers PE, Witte EV, Oshel JQ, Butler MS. Effects of Practical Blood Flow Restriction Training on Adolescent Lower-Body Strength. J Strength Cond Res. 2019 Oct;33(10):2674-2683. doi: 10.1519/JSC.0000000000002302. PMID 29084094
- [Result] Lu Y, Patel BH, Kym C, Nwachukwu BU, Beletksy A, Forsythe B, Chahla J. Perioperative Blood Flow Restriction Rehabilitation in Patients Undergoing ACL Reconstruction: A Systematic Review. Orthop J Sports Med. 2020 Mar 25;8(3):2325967120906822. doi: 10.1177/2325967120906822. eCollection 2020 Mar. PMID 32232065
- [Result] Weatherholt AM, Vanwye WR, Lohmann J, Owens JG. The Effect of Cuff Width for Determining Limb Occlusion Pressure: A Comparison of Blood Flow Restriction Devices. Int J Exerc Sci. 2019 Jan 1;12(3):136-143. doi: 10.70252/RWVU7100. eCollection 2019. PMID 30761200
- [Result] Ingram JG, Fields SK, Yard EE, Comstock RD. Epidemiology of knee injuries among boys and girls in US high school athletics. Am J Sports Med. 2008 Jun;36(6):1116-22. doi: 10.1177/0363546508314400. Epub 2008 Mar 28. PMID 18375784
- [Result] Powell JW, Barber-Foss KD. Injury patterns in selected high school sports: a review of the 1995-1997 seasons. J Athl Train. 1999 Jul;34(3):277-84. PMID 16558577
- [Result] Joseph AM, Collins CL, Henke NM, Yard EE, Fields SK, Comstock RD. A multisport epidemiologic comparison of anterior cruciate ligament injuries in high school athletics. J Athl Train. 2013 Nov-Dec;48(6):810-7. doi: 10.4085/1062-6050-48.6.03. Epub 2013 Oct 23. PMID 24143905
- [Result] Prue J, Roman DP, Giampetruzzi NG, Fredericks A, Lolic A, Crepeau A, Pace JL, Weaver AP. Side Effects and Patient Tolerance with the Use of Blood Flow Restriction Training after ACL Reconstruction in Adolescents: A Pilot Study. Int J Sports Phys Ther. 2022 Apr 2;17(3):347-354. doi: 10.26603/001c.32479. eCollection 2022. PMID 35391873

DOCUMENTS (1):
  • Informed Consent Form (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT05735236/ICF_002.pdf